CLINICAL TRIAL: NCT01416285
Title: The Impact of Heart Failure Center Program on The Progression of Biomarkers, Changes in Life Quality, Left Ventricular Ejection Fraction, and Cardiac Outcomes in Patients With Congestive Heart Failure
Brief Title: Impact of Heart Failure Center Program on Cardiac Outcomes in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, luck5748, Director of Heart Failure Research Center, Chang Gung Memorial Hospital
Other Study IDs: 98-1154B; CMRPG280251 (Other Grant/Funding Number: CHANG GUNG MEMORIAL HOSPITAL)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Death; Congestive Heart Failure
Keywords: Congestive heart failure (CHF); CHF education; self-care training; CHF center
MeSH Terms: conditions — Death; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At baseline and every 6-month visits, 3 ml of venous blood will be collected. At baseline and each 6-month visit, urinary albumin amount will be measured in the core lab in the hospital.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control group: control group receiving regular education from a nurse
- Case management group: This is the study group. Extensive education and case management program will be performed in this group.

SUMMARY:
Congestive heart failure (CHF) is a major public health problem worldwide. CHF carries a devastating prognosis, which resembles that of some types of malignant cancer. Despite substantial improvements in the management of the disease, the prognosis remains poor especially in advanced stages of the disease. For these patients, self-management plan includes monitoring of symptoms such as fatigue and shortness of breath, daily weighing, and knowing what to do if signs of deterioration appear, and when to report the changes to health. The investigators hypothesize that patients in the heart failure management programs that promote self-management by means of intensive education, edema index-assistance, and telephone follow-up can improve their functional status and quality of life, as well as the biomarkers of CHF, left ventricular systolic function, proteinuria and nutritional status.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is a major public health problem world-wide. CHF carries a devastating prognosis which resembles that of some types of malignant cancer. Its incidence rises steadily from 0.02 per 1000 population per year in those aged 25 to 34 years to 11.6 in those aged 85 years or older. Despite substantial improvements in the management of the disease, the prognosis remains poor especially in advanced stages of the disease. About half of the patients diagnosed with CHF die within 4 years of diagnosis. With the increasing number of patients with CHF being referred from hospital to primary health care, the demands for expanded services in primary health care have increased. Caring for patients with CHF often involves a number of physical, medical, behavioral, psychological and social factors, and requires appropriate attention to all aspects of care, both pharmacological and non-pharmacological. Educating patients about CHF treatment and the consequences of CHF has been shown to improve self-management behavior. For patients with CHF, the self-management plan includes monitoring of symptoms such as fatigue and shortness of breath, daily weighing, and knowing what to do if signs of deterioration appear, and when to report the changes to health care provider. In patients with CHF, the prognosis worsens considerably once malnutrition develops. Mortality at 18 months in unselected patients with CHF in whom cardiac cachexia had been diagnosed was as high as 50% compared to in non-cachectic patients from the same study population. In addition, amount of proteinuria has been known to be related to atherosclerosis burden and disease severity regarding lots of disease entities. The atherosclerosis score is also probably modifiable by life style intervention and educational program. CHF can also activate a few neurohormone and natriuretic peptides, among which brain natriuretic peptide is the most world-wide used. Summarized, in this study, to estimate the effect of CHF education and self-management program, the parameters adopted include blood brain natriuretic peptide and albumin levels, atherosclerosis scores, proteinuria, renal function, changes in life quality, left ventricular ejection fraction, and cardiac outcomes. In Taiwan, so far, the investigators don't have this kind of CHF education and self-care system. The investigators hypothesize that patients in the heart failure management programs that promote self-management by means of intensive education, edema index-assistance, and telephone follow-up can improve their functional status and quality of life, as well as the biomarkers of CHF, left ventricular systolic function, proteinuria and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. patients hospitalized due to acute cardiogenic pulmonary edema documented on chest x-ray and
2. left ventricular ejection fraction (LVEF) < 40% as documented by echocardiography; and
3. aged > 20 and < 80 years.

Exclusion Criteria:

1. the presence of systemic diseases such as hypothyroidism, decompensated liver cirrhosis, and systemic lupus erythematosus;
2. a disorder other than HF that might compromise survival within 6 months;
3. having implanted materials that could interfere with the bioimpedance analysis,
4. being bed-ridden for > 3 months and/or unable to stand alone;
5. having serum creatinine of > 5 mg/dl or nephritic syndrome;
6. having active cellulites, severe varicose veins, lymphedema or deep vein thrombosis over lower extremity;
7. undergoing dialysis within 2 weeks;
8. having severe coronary artery disease without complete revascularization therapy; and
9. being pregnant.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized due to acute cardiogenic pulmonary edema will be consecutively enrolled in the HF center of Chang Gung Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-05-30 (Actual); Study Completion 2012-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CHAO-HUNG WANG, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jaarsma T, van der Wal MH, Lesman-Leegte I, Luttik ML, Hogenhuis J, Veeger NJ, Sanderman R, Hoes AW, van Gilst WH, Lok DJ, Dunselman PH, Tijssen JG, Hillege HL, van Veldhuisen DJ; Coordinating Study Evaluating Outcomes of Advising and Counseling in Heart Failure (COACH) Investigators. Effect of moderate or intensive disease management program on outcome in patients with heart failure: Coordinating Study Evaluating Outcomes of Advising and Counseling in Heart Failure (COACH). Arch Intern Med. 2008 Feb 11;168(3):316-24. doi: 10.1001/archinternmed.2007.83. PMID 18268174
- [Result] Hoekstra T, Lesman-Leegte I, van der Wal M, Luttik ML, Jaarsma T. Nurse-led interventions in heart failure care: patient and nurse perspectives. Eur J Cardiovasc Nurs. 2010 Dec;9(4):226-32. doi: 10.1016/j.ejcnurse.2010.01.006. Epub 2010 Mar 4. PMID 20202912
- [Result] Riegel B, Lee CS, Dickson VV; Medscape. Self care in patients with chronic heart failure. Nat Rev Cardiol. 2011 Jul 19;8(11):644-54. doi: 10.1038/nrcardio.2011.95. PMID 21769111
- [Derived] Mao CT, Liu MH, Hsu KH, Fu TC, Wang JS, Huang YY, Yang NI, Wang CH. Effect of multidisciplinary disease management for hospitalized heart failure under a national health insurance programme. J Cardiovasc Med (Hagerstown). 2015 Sep;16(9):616-24. doi: 10.2459/JCM.0000000000000089. PMID 25105284
- [Derived] Liu MH, Wang CH, Huang YY, Tung TH, Lee CM, Yang NI, Liu PC, Cherng WJ. Edema index established by a segmental multifrequency bioelectrical impedance analysis provides prognostic value in acute heart failure. J Cardiovasc Med (Hagerstown). 2012 May;13(5):299-306. doi: 10.2459/JCM.0b013e328351677f. PMID 22367574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled patients consecutively hospitalized for acute or decompensated chronic heart failure in the heart failure center of Chang Gung Memorial Hospital, Keelung, Taiwan from June 1, 2010 to May 30, 2012.
Pre-assignment Details: Of 470 enrolled participants, 121 were excluded (42 were excluded because of met exclusion criteria, 42 refused to participate, and 26 were excluded because of other reasons) , 349 met inclusion criteria and randomized to into the control and the case management groups.
Period: Overall Study
Arm/Group | Control Group | Case Management Group
Started | 175 | 174
Completed | 175 | 165
Not Completed | 0 | 9
Not completed — owing to the care model or moving to other cities of the country | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Case Management Group | Total
Number analyzed (Participants) | 175 | 174 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12.6) | 59.2 (13.6) | 60.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 47 | 105
  Male | 117 | 127 | 244
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Previous hospitalization due to Heart Failure [Count of Participants; unit: Participants] | 70 | 55 | 125
New York Heart Association functional class [Count of Participants; unit: Participants] — Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
  Participants
    II | 34 | 34 | 68
    III | 130 | 134 | 264
    IV | 11 | 6 | 17
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage of blood ejected] | 35.1 (14.3) | 36.9 (15.8) | 36.0 (15.1)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 122.9 (21.9) | 123 (18.2) | 122.9 (20.1)
  Diastolic | 73.4 (14.3) | 75.3 (12.3) | 74.3 (13.4)
Co-morbidity [Count of Participants; unit: Participants]
  Diabetes mellitus | 82 | 66 | 148
  Chronic Kidney Disease | 49 | 42 | 91
  Hypertension | 116 | 110 | 226
  Atrial Fibrillation | 49 | 47 | 96
  Chronic Obstructive Pulmonary Disease | 17 | 21 | 38
Cause [Count of Participants; unit: Participants]
  Ischemic | 85 | 91 | 176
  Valvular | 27 | 23 | 50
  Idiopathic | 36 | 29 | 65
  Living alone | 58 | 56 | 114
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (5.7) | 25.1 (5) | 25.2 (5.4)
Medication [Count of Participants; unit: Participants]
  Angiotensin-Converting Enzyme Inhibitor or Angiotensin Receptor Blocker | 140 | 135 | 275
  Beta-Blocker | 78 | 81 | 159
  Digoxin | 49 | 49 | 98
  Diuretic | 112 | 94 | 206
Laboratory values [Mean (Standard Deviation); unit: g/dl]
  Hemoglobin | 13.3 (2.1) | 13.7 (2) | 13.5 (3.6)
  Albumin | 3.5 (0.5) | 3.6 (0.5) | 3.6 (0.5)
Heart rate [Mean (Standard Deviation); unit: beats/min] | 79.7 (14.7) | 77.7 (11.7) | 78.7 (13.3)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 69.1 (36.1) | 74.7 (23.8) | 71.8 (30.6)
B-type natriuretic peptide [Mean (Standard Deviation); unit: pg/ml] | 637 (756) | 653 (738) | 646 (742)
Serum sodium [Mean (Standard Deviation); unit: mEq/l] | 138.6 (3.4) | 138.9 (3.8) | 138.7 (3.6)
Total bilirubin [Mean (Standard Deviation); unit: mg/dl] | 1.1 (0.6) | 1.1 (0.7) | 1.1 (0.7)
QRS complex [Mean (Standard Deviation); unit: msec] | 102.2 (26.6) | 103.5 (25.1) | 102.9 (24.5)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Death, Heart Failure-related Re-hospitalizations, and a Composite Outcome of Both Death and Heart Failure-related Re-hospitalizations
Description: Follow-up began after randomization. Follow-up data were prospectively obtained every month from hospital records, personal communication with patients' physicians, telephone interviews, and records of regular visits to staff physicians' outpatient clinics. 'Re-hospitalization'was defined as heart failure-related re-hospitalization.'All causes of death' was also considered to be an event. All-cause death was chosen as an endpoint because of the inter-relationship of heart failure with many other comorbidities in the patient cohort. A committee of three cardiologists adjudicated all hospitalizations without knowledge of the patients' clinical data to determine whether events were related to worsening heart failure. Based on these two different endpoints, time to the first event was analyzed.
Time Frame: 2 year
Population: Death, HF-related rehospitalization, and composite of death and HF-related rehospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Case Management Group
Number analyzed (Participants) | 175 | 165
Participants
  Death | 36 | 15
  Heart Failure-related re-hospitalization | 41 | 18
  Death and Heart Failure-related re-hospitalization | 63 | 28
Statistical Analysis 1: Comparison: Control Group vs Case Management Group; All-cause death; Test type: Superiority; p = 0.004, Kaplan-Meier and COX regression; Univariate and multi-variable
Statistical Analysis 2: Comparison: Control Group vs Case Management Group; Heart failure-related re-hospitalizations; Test type: Superiority; p = 0.003, Kaplan-Meier and COX regression; Univariate and multi-variable
Statistical Analysis 3: Comparison: Control Group vs Case Management Group; a composite outcome of both death and heart failure-related re-hospitalizations; Test type: Superiority; p < 0.001, Kaplan-Meier and COX regression; Univariate and multi-variable

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Control Group | Case Management Group
All-Cause Mortality (participants affected / at risk) | 36/175 | 15/165
Serious Adverse Events (participants affected / at risk) | 41/175 | 18/165
Other Adverse Events (participants affected / at risk) | 0/175 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=175) | Case Management Group (N=165)
Heart failure-related re-hospitalizations (Cardiac disorders) | 41 (41) | 18 (18) — Patients were re-hospitalized due to unanticipated worsening of heart failure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No